CLINICAL TRIAL: NCT03173235
Title: Plasma Concentrations of Calcium, Phosphate, FGF23, Klotho, 25 (OH) D3 and 1,25 (OH) 2D3 from Patients Who Wants to Have Children
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Vitamin D
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infertile women: Women which desire to have children but are probable infertile between 18 and 45 year old
  Interventions: Diagnostic Test: Plasma level of vitamin D
- healthy women: Healthy women without systemic diseases in the age of 18 to 45 years
  Interventions: Diagnostic Test: Plasma level of vitamin D

INTERVENTIONS:
Diagnostic Test: Plasma level of vitamin D — messurement of plasma level of vitamin D

SUMMARY:
1,25-dihydroxy-vitamin D3 (1,25 (OH) 2D3) or calcitriol regulates plasma calcium and phosphate concentrations in the blood by stimulating intestinal absorption and renal reabsorption of calcium and phosphate. 1.25 (OH) 2D3 is formed by the renal 1α25OH vitamin D-hydroxylase (Cyp27b1) and inactivated by the renal 25-hydroxy vitamin D-24-hydroxylase (Cyp24). Unpublished studies in mice revealed an inhibitory effect of 1.25 (OH) 2D3 on embryo implanation. An excess of 1.25 (OH) 2D3 could therefore lead to female infertility. The excess of 1.25 (OH) 2D3 could result from uncritical vitamin D intake with insufficient negative feedback by FGF23 / Klotho. The aim of the study is to identify patients with an excess of 1.25 (OH) 2D3.

DETAILED DESCRIPTION:
The physiological institute of the University Tübinge has succeeded in preventing vascular calcification in Klotho-deficient mice by inhibiting osteogenic signal transduction. The animals reach an almost normal life span despite increased 1.25 (OH) 2D3, Ca2 + and phosphate plasma concentrations. The male animals are again fertilized, but not the female animals. However, if the plasma concentrations of 1.25 (OH) 2D3 are normalized by administration of a vitamin-poor diet, the female animals are fertilized within two weeks. Further investigations revealed an inhibitory effect of 1.25 (OH) 2D3 on the implantation of the embryo. In the meantime the 1,25 (OH) 2D3-dependent signal transduction could be revealed, which prevents the implantation of the embryo. The vitamin D receptor and the elements of signal transduction are also expressed in the human endometrium. It is therefore possible that increased 1.25 (OH) 2D3 plasma concentrations also prevent embryo implantation in humans.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Known systemic diseases, e.g. Autoimmune disease, scleroderma, malignant disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women in the age of 18 to 45 years
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Plasma level of 25(OH)D3 and 1,25(OH)2D3 | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University Women's Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No